CLINICAL TRIAL: NCT00109707
Title: A Phase IA/II Multicenter, Dose-escalation Study of Oral AMN107 on a Continuous Daily Dosing Schedule in Adult Patients With Imatinib-resistant/Intolerant CML in Chronic or Accelerated Phase or Blast Crisis, Relapsed/Refractory Ph+ ALL, and Other Hematologic Malignancies.
Brief Title: A Study of Oral AMN107 in Adults With Chronic Myelogenous Leukemia (CML) or Other Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2101
Record Dates: First submitted 2005-05-02; First posted 2005-05-03 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Chronic Myelogenous Leukemia; Acute Lymphoblastic Leukemia (Philadelphia Chromosome Positive); Hypereosinophilic Syndrome; Systemic Mastocytosis
Keywords: CML in blast crisis; CML in chronic phase; CML in accelerated phase; Gleevec resistance; Gleevec intolerant; Gleevec and CML; imatinib resistance; imatinib intolerant; Hypereosinophilic Syndrome; Systemic Mastocytosis; Chronic eosinophilic syndrome; Philadelphia chromosome positive acute lymphoblastic leukemia; HES; CEL; CML; SM; Ph+ ALL refractory to standard therapy; Ph+ALL relapsed; AMN107A
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hypereosinophilic Syndrome; Mastocytosis, Systemic | interventions — nilotinib

ARMS (3):
- CML-CP With Prior Imatinib Only (Experimental): Imatinib-resistant / intolerant PH+ CML-CP patients
  Interventions: Drug: Nilotinib
- CML-AP With Prior Imatinib Onl (Experimental): Imatinib-resistant / intolerant PH+ CML-AP patients
  Interventions: Drug: Nilotinib
- CML-CP (Experimental): Imatinib-resistant / intolerant PH+ CML-CP patients
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib

SUMMARY:
The purpose of this trial is to assess the efficacy, safety, tolerability, biologic activity, and pharmacokinetics of AMN107 in six groups of patients with one of the following conditions:

Relapsed/refractory Ph+ Acute lymphoblastic leukemia (ALL) (arm 1)

Group A - Imatinib failure only (arms 2, 3 and 4)

* imatinib-resistant or intolerant CML - Chronic Phase (CP)
* imatinib-resistant or intolerant CML - Accelerated Phase (AP)
* imatinib-resistant or intolerant CML - Blast Crisis (BC)

Group B - Imatinib and other TKI failure (arms 2, 3 and 4)

* imatinib-resistant or intolerant CML - Chronic Phase (CP)
* imatinib-resistant or intolerant CML - Accelerated Phase (AP)
* imatinib-resistant or intolerant CML - Blast Crisis (BC)

Hypereosinophilic syndrome/chronic eosinophilic leukemia (HES/CEL) (arm 5)

Systemic mastocytosis (Sm) (arm 6)

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria include:

* Patients with CML in blast crisis, CML in accelerated phase defined as never in blast crisis phase, or CML in chronic phase defined as never been in blast crisis phase or accelerated phase who have: *developed progressive disease during therapy with at least 600 mg of imatinib per day, -OR- *patients with CML on imatinib therapy, at any dose, developing progressive disease and the presence of a genetic mutation likely to result in imatinib resistance -OR- *have developed an intolerance to imatinib
* Relapsed or refractory Ph+ ALL
* Hypereosinophilic syndrome/chronic eosinophilic leukemia.
* Systemic mastocytosis who have a clinical indication for treatment.
* Prior imatinib therapy for patients with Ph+ ALL, HES/CEL and SM is permitted but is not required
* CML patients who have been treated with an investigational tyrosine kinase inhibitor who otherwise meet the definition of imatinib-resistance or intolerance are eligible
* Written informed consent prior to any study procedures being performed

Exclusion Criteria:

* Impaired cardiac function
* Patients with severe/chronic or uncontrolled medical conditions (including but not limited to diabetes, infections, GI impairment, CNS infiltration, liver and kidney disease)
* Prior and concomitant use of certain medications (including but not limited to warfarin, chemotherapy, hematopoietic colony-stimulating growth factors, medications that can affect electrocardiogram test results, other investigational drugs )
* Women who are pregnant or breastfeeding
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients unwilling to comply with the protocol.
* Known diagnosis of human immunodeficiency virus (HIV) infection

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticlas, Study Director — Novartis Pharmaceuticals
Locations (95):
- United States (24):
  - City of Hope National Medical Center, Duarte, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute Dept.of H. Lee Moffitt, Tampa, Florida
  - University of Chicago Medical Center Dept. of U. of Chicago Hosp(3), Chicago, Illinois
  - University of Illinois at Chicago Divisionof Hematology/Oncology, Chicago, Illinois
  - Indiana Blood and Marrow Institute Dept of Indiana Blood&Mar (2), Beech Grove, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center/Johns Hopkins Med. Div.of Hematologic Malignancie, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System Clinical Trials Office, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute Rosewell SC, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - The Jones Clinic, Germantown, Tennessee
  - Vanderbilt University Medical Center, Clinical Trials Center Investigational Drug Services, Nashville, Tennessee
  - MD Anderson Cancer Center/University of Texas, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Australia (3):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Prahran, Victoria
- Novartis Investigative Site, Vienna, Austria
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Haine-Saint-Paul
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Yvoir
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Vejle, Denmark
- Novartis Investigative Site, HUS Helsinki, Finland
- France (10):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (8):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt/M
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
- Novartis Investigative Site, Pokfulam, Hong Kong, Hong Kong
- Italy (11):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Napoli
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Grafton, Auckland, New Zealand
- Novartis Investigative Site, Oslo, Norway
- Poland (4):
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Hwasun-gun, Jeollanam-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Taegu
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Uppsala
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Geneva
- Novartis Investigative Site, Niaosong Township, Taiwan, Taiwan
- United Kingdom (7):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Glasgow - Scotland
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Hochhaus A, Baccarani M, Giles FJ, le Coutre PD, Muller MC, Reiter A, Santanastasio H, Leung M, Novick S, Kantarjian HM. Nilotinib in patients with systemic mastocytosis: analysis of the phase 2, open-label, single-arm nilotinib registration study. J Cancer Res Clin Oncol. 2015 Nov;141(11):2047-60. doi: 10.1007/s00432-015-1988-0. Epub 2015 May 23. PMID 26002753
- [Derived] Hochhaus A, le Coutre PD, Kantarjian HM, Baccarani M, Erben P, Reiter A, McCulloch T, Fan X, Novick S, Giles FJ. Effect of the tyrosine kinase inhibitor nilotinib in patients with hypereosinophilic syndrome/chronic eosinophilic leukemia: analysis of the phase 2, open-label, single-arm A2101 study. J Cancer Res Clin Oncol. 2013 Dec;139(12):1985-93. doi: 10.1007/s00432-013-1529-7. Epub 2013 Sep 22. PMID 24057647
- [Derived] Stein AM, Martinelli G, Hughes TP, Muller MC, Beppu L, Gottardi E, Branford S, Soverini S, Woodman RC, Hochhaus A, Kim DW, Saglio G, Radich JP. Rapid initial decline in BCR-ABL1 is associated with superior responses to second-line nilotinib in patients with chronic-phase chronic myeloid leukemia. BMC Cancer. 2013 Apr 2;13:173. doi: 10.1186/1471-2407-13-173. PMID 23547655
- [Derived] Kantarjian HM, Giles FJ, Bhalla KN, Pinilla-Ibarz J, Larson RA, Gattermann N, Ottmann OG, Hochhaus A, Radich JP, Saglio G, Hughes TP, Martinelli G, Kim DW, Shou Y, Gallagher NJ, Blakesley R, Baccarani M, Cortes J, le Coutre PD. Nilotinib is effective in patients with chronic myeloid leukemia in chronic phase after imatinib resistance or intolerance: 24-month follow-up results. Blood. 2011 Jan 27;117(4):1141-5. doi: 10.1182/blood-2010-03-277152. Epub 2010 Nov 22. PMID 21098399
- [Derived] Kantarjian HM, Giles F, Gattermann N, Bhalla K, Alimena G, Palandri F, Ossenkoppele GJ, Nicolini FE, O'Brien SG, Litzow M, Bhatia R, Cervantes F, Haque A, Shou Y, Resta DJ, Weitzman A, Hochhaus A, le Coutre P. Nilotinib (formerly AMN107), a highly selective BCR-ABL tyrosine kinase inhibitor, is effective in patients with Philadelphia chromosome-positive chronic myelogenous leukemia in chronic phase following imatinib resistance and intolerance. Blood. 2007 Nov 15;110(10):3540-6. doi: 10.1182/blood-2007-03-080689. Epub 2007 Aug 22. PMID 17715389
- [Derived] Kantarjian H, Giles F, Wunderle L, Bhalla K, O'Brien S, Wassmann B, Tanaka C, Manley P, Rae P, Mietlowski W, Bochinski K, Hochhaus A, Griffin JD, Hoelzer D, Albitar M, Dugan M, Cortes J, Alland L, Ottmann OG. Nilotinib in imatinib-resistant CML and Philadelphia chromosome-positive ALL. N Engl J Med. 2006 Jun 15;354(24):2542-51. doi: 10.1056/NEJMoa055104. PMID 16775235
- See also: Results for CAMN107A2101 on the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 100 centers in 22 countries.
Pre-assignment Details: A total of 507 participants were randomized in the core study, out of which 136 participants entered the extension study.
Groups:
- CML-CP With Prior Imatinib Only: Adult participants PH+ CML-CP ( Chronic Phase Chronic Myeloid Leukemia) without prior TKI treatment with either resistant / intolerant to Imatinib received 400 mg Nilotinib orally twice daily up to the end of treatment (September-2012).
- CML-AP With Prior Imatinib Only: Adult participants PH+ CML-AP (Accelerated Phase Chronic Myeloid Leukemia) without prior TKI treatment with either resistant / intolerant to Imatinib received 400 mg Nilotinib orally twice daily up to the end of treatment (September-2012).
- CML-CP: Adult participants PH+ CML-CP in addition to prior TKI treatment with either resistant / intolerant to Imatinib received 400 mg Nilotinib orally twice daily up to the end of treatment (September-2012).
Period: Overall Study
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only | CML-CP
Started | 321 | 137 | 49
Entered Extension Study | 106 | 15 | 15
Completed | 67 | 8 | 8
Not Completed | 254 | 129 | 41
Not completed — Discontinued in core study without entering the extension study | 215 | 122 | 34
Not completed — Abnormal laboratory values | 1 | 0 | 0
Not completed — Administrative problems | 2 | 0 | 1
Not completed — Adverse Event | 10 | 2 | 3
Not completed — Death | 4 | 0 | 0
Not completed — Disease progression | 12 | 4 | 3
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Patient withdrew consent | 6 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CML-CP With Prior Imatinib Only: Adult participants PH+ CML-CP without prior TKI treatment with either resistant / intolerant to Imatinib received 400 mg Nilotinib orally twice daily up to the end of treatment (September-2012).
- CML-AP With Prior Imatinib Only: Adult participants PH+ CML-AP without prior TKI treatment with either resistant / intolerant to Imatinib received 400 mg Nilotinib orally twice daily up to the end of treatment (September-2012).
- Total: Total of all reporting groups
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only | CML-CP | Total
Number analyzed (Participants) | 321 | 137 | 49 | 507
Age, Customized [Count of Participants; unit: Participants]
  <35 years | 22 | 8 | 3 | 33
  ≥35 to <55 years | 104 | 49 | 16 | 169
  ≥55 to <65 years | 97 | 39 | 12 | 148
  ≥65 years | 98 | 41 | 18 | 157
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 61 | 25 | 245
  Male | 162 | 76 | 24 | 262

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Cytogenetic Response (MCyR)
Description: Major Cytogenetic Response (MCyR) is defined as Complete Cytogenetic Response (CCyR: 0% Ph-chromosome-positive cells in metaphase in bone marrow) or Partial Cytogenetic Response (PCyR: 1-35% Ph-chromosome-positive cells in metaphase in bone marrow).
Time Frame: Up to End of the Treatment (Approximately 7.5 years)
Population: Full Analysis Set (FAS): All participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only | CML-CP
Number analyzed (Participants) | 321 | 137 | 49
Participants | 191 | 44 | 22

2. Primary Outcome: Number of Participants Confirmed Overall Hematological Response (Phase II)
Description: Hematologic response is defined as the percentage of participants in complete hematologic response (defined as the following present for at least 4 weeks: WBC count <10 x 109/L, Platelet count <450 x 109/L, Basophils <5%, No blasts and promyelocytes in peripheral blood, Myelocytes + metamyelocytes < 5% in peripheral blood, No evidence of extramedullary disease, including spleen and liver).
  Hematological response was a primary outcome measure for Arm CML-AP with prior imatinib only.
Time Frame: Up to End of the Treatment (Approximately 7.5 years)
Population: Full Analysis Set (FAS): All participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CML-AP With Prior Imatinib Only
Number analyzed (Participants) | 137
Participants | 76

3. Secondary Outcome: Number of Participants With Overall Major Cytogenetic Responses (Phase II)
Description: Cytogenetic responses (CyRs) in CML are based on the percentage of Ph+ metaphases in bone marrow; a value of 0% Ph+ metaphases defines a complete cytogenetic response (CCyR) and >0% to 35% defines a major cytogenetic response (MCyR). Achievement of CCyR is associated with a significant survival advantage in participants with CML-CP. MCyR was categorized as either CCyR or partial cytogenetic response (PCyR).
Time Frame: Up to End of the Treatment (Approximately 7.5 years)
Population: Full Analysis Set (FAS): All participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only | CML-CP
Number analyzed (Participants) | 321 | 137 | 49
participants | 191 | 44 | 22

4. Secondary Outcome: Number of Participants With Complete Hematologic Response (Phase II)
Description: A Complete Hematologic Response (CHR) is obtained when all the following criteria are met: WBC ≤ institutional ULN; platelets ≤ 450,000/mm3; ≤20% basophils in peripheral blood; no blasts or promyelocytes in PB cells; < 5% myelocytes plus metamyelocytes in PB cells; no extra-medullary involvement including no hepatomegaly or splenomegaly.
Time Frame: Up to End of the Treatment (Approximately 7.5 years)
Population: Full Analysis Set (FAS): All participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only | CML-CP
Number analyzed (Participants) | 321 | 137 | 35
participants | 158 | 76 | 27

5. Secondary Outcome: Participants With (MMR) Major Molecular Response (Phase II)
Description: MMR was defined for participants who demonstrated a reduction in BCR-ABL/control gene % transcripts to ≤0.1% based on international scale. The control gene used may have been either BCR or ABL.
Time Frame: Up to End of the Treatment (Approximately 7.5 years)
Population: Full Analysis Set (FAS): All participants who received at least one dose of study medication.
  Major molecular response was not an efficacy variable for participants who received the CML-CP with prior imatinib and other TKI (Group B E8)
Measure: Count of Participants; unit: Participants
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only
Number analyzed (Participants) | 299 | 122
Participants | 106 | 18

6. Secondary Outcome: Time to Progression (TTP) (Phase II)
Description: Time to Progression was defined as the time from the start of nilotinib to the earliest date of Disease Progression (PD), discontinuation due to PD or death.
  Disease progression was defined as an increase in the number of circulating leukemic cells via cytogenetic assessment using real-time quantitative reverse transcriptase polymerase chain reaction (PCR).
Time Frame: Up to End of the Treatment (Approximately 7.5 years)
Population: Full Analysis Set (FAS): All participants who received at least one dose of study medication.
  Time to progression was not an efficacy variable for participants who received the CML-CP with prior imatinib and other TKI (Group B E8).
Measure: Median (Full Range); unit: Months
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only
Number analyzed (Participants) | 321 | 137
Months | 55.6 [0.1 to 77.8] | 15.9 [0.1 to 75.7]

7. Secondary Outcome: Overall Survival (OS) (Phase II)
Description: OS was calculated for all participants as the time between the start of nilotinib and death. Participants were followed for survival after discontinuation, every 3 months, and were included in the analysis of OS. Censoring was at the date of the last contact for discontinued participants and followed up for survival.
Time Frame: Up to End of the Treatment (Approximately 7.5 years)
Population: Full Analysis Set (FAS): All participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only | CML-CP
Number analyzed (Participants) | 321 | 137 | 49
months | NA [77.93 to NA] — Median OS was not reached as there were an insufficient number of participants | 47.54 [38.24 to 64.30] | NA [NA to NA] — Median OS was not reached as there were an insufficient number of participants

8. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events to Evaluate Long Term Safety
Description: Adverse events (AEs) were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: From First Participant First Visit to Last Participant Last Visit (Approximately 7.5 years)
Population: Safety set: All participants who received at least one dose of study medication and had at least one post baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only | CML-CP
Number analyzed (Participants) | 321 | 137 | 49
Participants
  Serious Adverse Events | 61 | 26 | 5
  Adverse Events | 57 | 17 | 7

ADVERSE EVENTS:
Time Frame: From First Participant First Visit to Last Participant Last Visit (Approximately 7.5 years)
Description: Safety set: All participants who received at least one dose of study medication and had at least one post baseline safety assessment.
Arm/Group | CML-CP With Prior Imatinib Only | CML-AP With Prior Imatinib Only | CML-CP
All-Cause Mortality (participants affected / at risk) | 13/321 | 14/137 | 0/49
Serious Adverse Events (participants affected / at risk) | 146/321 | 55/137 | 21/49
Other Adverse Events (participants affected / at risk) | 319/321 | 136/137 | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CML-CP With Prior Imatinib Only (N=321) | CML-AP With Prior Imatinib Only (N=137) | CML-CP (N=49)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 11 | 3
Neutropenia (Blood and lymphatic system disorders) | 7 | 8 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 2
Angina pectoris (Cardiac disorders) | 12 | 0 | 0
Myocardial infarction (Cardiac disorders) | 7 | 5 | 0
Acute myocardial infarction (Cardiac disorders) | 6 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 0 | 1
Coronary artery disease (Cardiac disorders) | 5 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 2 | 0 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 0
Catarac (Eye disorders) | 2 | 0 | 0
Diplopia (Eye disorders) | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 6 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Pyrexia (General disorders) | 9 | 6 | 2
Chest pain (General disorders) | 4 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 4 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Peritonitis (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 7 | 4
Sepsis (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 0
Lipase increased (Investigations) | 3 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Back pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 0
Brain oedema (Nervous system disorders) | 2 | 0 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Haematoma (Vascular disorders) | 2 | 0 | 1
Temporal arteritis (Vascular disorders) | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 3 | 1
Aphasia (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CML-CP With Prior Imatinib Only (N=321) | CML-AP With Prior Imatinib Only (N=137) | CML-CP (N=49)
Thrombocytopenia (Blood and lymphatic system disorders) | 107 | 60 | 16
Anaemia (Blood and lymphatic system disorders) | 71 | 61 | 9
Neutropenia (Blood and lymphatic system disorders) | 57 | 39 | 15
Leukopenia (Blood and lymphatic system disorders) | 16 | 11 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 16 | 0 | 0
Conjunctivitis (Eye disorders) | 20 | 0 | 0
Nausea (Gastrointestinal disorders) | 121 | 41 | 13
Diarrhoea (Gastrointestinal disorders) | 93 | 34 | 6
Vomiting (Gastrointestinal disorders) | 92 | 30 | 7
Constipation (Gastrointestinal disorders) | 88 | 31 | 10
Abdominal pain (Gastrointestinal disorders) | 47 | 17 | 8
Abdominal pain upper (Gastrointestinal disorders) | 46 | 21 | 6
Dyspepsia (Gastrointestinal disorders) | 33 | 0 | 7
Fatigue (General disorders) | 105 | 28 | 13
Pyrexia (General disorders) | 66 | 49 | 8
Oedema peripheral (General disorders) | 55 | 27 | 5
Asthenia (General disorders) | 53 | 24 | 12
Chest pain (General disorders) | 19 | 0 | 4
Pain (General disorders) | 19 | 10 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 32 | 10 | 0
Nasopharyngitis (Infections and infestations) | 80 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 41 | 7 | 5
Urinary tract infection (Infections and infestations) | 28 | 0 | 4
Bronchitis (Infections and infestations) | 26 | 0 | 4
Sinusitis (Infections and infestations) | 22 | 0 | 5
Influenza (Infections and infestations) | 21 | 0 | 0
Rhinitis (Infections and infestations) | 16 | 0 | 3
Procedural pain (Injury, poisoning and procedural complications) | 17 | 0 | 0
Lipase increased (Investigations) | 55 | 8 | 10
Alanine aminotransferase increased (Investigations) | 39 | 14 | 8
Weight decreased (Investigations) | 30 | 15 | 2
Blood bilirubin increased (Investigations) | 29 | 14 | 4
Aspartate aminotransferase increased (Investigations) | 24 | 7 | 5
Blood creatine phosphokinase increased (Investigations) | 19 | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 19 | 0 | 0
Amylase increased (Investigations) | 18 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 50 | 12 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 27 | 12 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 22 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 22 | 10 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 | 10 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 17 | 15 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 86 | 20 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 63 | 0 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 63 | 18 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 60 | 19 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 45 | 9 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 43 | 14 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 32 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 16 | 0 | 3
Headache (Nervous system disorders) | 114 | 0 | 11
Dizziness (Nervous system disorders) | 35 | 0 | 5
Paraesthesia (Nervous system disorders) | 17 | 0 | 0
Insomnia (Psychiatric disorders) | 40 | 0 | 2
Depression (Psychiatric disorders) | 28 | 0 | 3
Anxiety (Psychiatric disorders) | 20 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 17 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 91 | 21 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 | 14 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 39 | 16 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 21 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 17 | 2
Rash (Skin and subcutaneous tissue disorders) | 118 | 39 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 104 | 18 | 9
Night sweats (Skin and subcutaneous tissue disorders) | 37 | 7 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 36 | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 34 | 8 | 1
Erythema (Skin and subcutaneous tissue disorders) | 30 | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 26 | 7 | 3
Skin lesion (Respiratory, thoracic and mediastinal disorders) | 19 | 0 | 3
Hypertension (Vascular disorders) | 37 | 0 | 5
Tachycardia (Cardiac disorders) | 0 | 7 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 7 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 7 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 9 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 14 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 7 | 3
Chills (General disorders) | 0 | 15 | 1
Pneumonia (Infections and infestations) | 0 | 7 | 3
White blood cell count decreased (Investigations) | 0 | 11 | 0
Haemoglobin decreased (Investigations) | 0 | 9 | 0
Haemoglobin decreased (Investigations) | 0 | 7 | 0
Platelet count decreased (Investigations) | 0 | 7 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 7 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 9 | 0
Haematoma (Vascular disorders) | 0 | 10 | 0
Hypotension (Vascular disorders) | 0 | 10 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 3
Inflammation (General disorders) | 0 | 0 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 0 | 8
Herpes simplex (Infections and infestations) | 0 | 0 | 3
Herpes zoster (Infections and infestations) | 0 | 0 | 3
Periodontitis (Infections and infestations) | 0 | 0 | 3
Weight increased (Investigations) | 0 | 0 | 5
Blood glucose increased (Investigations) | 0 | 0 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.